CLINICAL TRIAL: NCT06771752
Title: Adherence to 24-Hour Movement Guidelines and Association With Diet Quality in Multi-Disciplinary Football Team Staff
Status: Completed | Type: Observational
Sponsor: University Ramon Llull (Other)
Responsible Party: Principal Investigator, Blanca Roman-Viñas, MD, Professor of Sports Medicine, University Ramon Llull
Other Study IDs: 2024-12-02
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity; Diet Quality; Staff; Soccer
Keywords: 24 hour movement; diet quality; football; physical activity; nutrition; strength training; football staff; soccer; soccer staff
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multidisciplinary Football Staff
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The questionnaire will be made comprised of the questions taken from the Whole Day Matters Toolkit (WDMT) 24-hour movement questionnaire (The Canadian Society for Exercise Physiology, 2021), which is based on the official 24-hour movement guidelines (Ross et al., 2020) (see appendix). For diet quality, Mini-EAT, a short dietary screening tool will be used (Lara-Breitinger et al., 2023) (see appendix). The questionnaire will be open for two months during the football mid-season time period (January 15th to March 15th). The principal investigator will distribute the questionnaire digitally via Google Forms. It will be sent directly to sports staff professionals, individually and to football clubs and to universities to distribute to their cohort. Only people with the link will be able to access the questionnaire. Participants will answer the questionnaire, which will take roughly 10 minutes, completing the intervention.
  Other Names: Whole Day Matters Toolkit: 24-hour movement questionnaire by The Canadian Society for Exercise Physiology; Mini-Eat dietary questionnaire

SUMMARY:
The goal of this observational study is to assess whether adherence to 24-hour movement guidelines is associated with diet quality in professional football staff, an underrepresented population affected by irregular schedules, travel, and high-pressure environments. The main objectives are to:

* Assess and describe the sleep quality of football sports staff
* Measure and contextualise the adherence to 24-hour movement guidelines in football sports staff
* Analyse and describe the diet quality of football sports staff
* Describe correlations between job title, gender and location for physical movement and diet quality

Participants will answer a questionnaire that incorporates:

* Personal descriptives (height, weight, age, location, job title)
* Data on physical activity (movement, sleep, sedentary behaviour, strength training, screen time) based on the Canadian 24-hour Movement Guidelines
* The Mini-EAT dietary screening tool that evaluates diet quality (intake of fruits, vegetables, whole grains, dairy, and sweets)

Statistical analyses will examine adherence levels, diet quality and the potential associations, aiming at informing health and performance strategies for football staff.

DETAILED DESCRIPTION:
This study investigates the relationship between adherence to 24-hour movement guidelines and diet quality among professional football sports staff, addressing the challenges posed by irregular schedules, travel and high-pressure environments. The aim is to determine whether staff meet the health recommendations they advocate for players and to inform strategies that enhance their health and performance. Using an observational and cross-sectional research design, the study will collect data on physical activity according to the Canadian 24-hour Movement Guidelines to assess adherence, and the validated Mini-EAT dietary screening tool to evaluate diet quality. The dependent variables include factors such as physical activity levels moderate-to-vigorous physical activity (MVPA), light physical activity (LPA), sedentary time, sleep quality and consistency, strength training, sedentary breaks, and screen time usage. Diet quality is assessed through the frequency of intake of various food groups (e.g., fruits, vegetables, legumes, whole grains, dairy, and sweets) and summarised with an overall diet quality score. There is a minimum of 229 participants required and the questionnaire will be distributed to individuals with confirmed employment of football staff, football clubs and universities with football teams. Statistical analyses will include descriptive statistics to summarise participant characteristics, adherence levels, and diet quality scores, MANOVA, Shapiro-Wilk to assess normality, with Pearson's or Spearman's correlations (depending on normality distribution) to examine associations between adherence scores and diet quality. Chi-square tests will identify relationships between categorical adherence levels and diet quality. These findings will inform targeted interventions to improve health outcomes for football staff, enabling them to better support players while maintaining their own performance. The proposed start date of the study is January 2025.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who work in football / soccer in professional leagues or semi-professional leagues in both men's and women's teams
* Individuals aged between 18 and 65
* Individuals who have confirmed status of their occupation on LinkedIn or football club website

Exclusion Criteria:

* Jobs in other sports besides football / soccer
* No public profile on LinkedIn or football club website to confirm job status
* No signing of the consent form in the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of professional football sports staff, including roles such as:
  * Manager / Head Coach
  * Assistant Coach
  * Goalkeeping Coach
  * Strength and Conditioning Coach
  * Talent Scout
  * Player Development Coach
  * Performance Coach
  * Sports Scientist
  * Performance Nutritionist
  * Sports Psychologist
  * Physical Therapist
  * Performance Analyst
  * Team Doctor
  * Physiotherapist
  * Performance Chef
  * Referee
  The study population will not be limited to one country or location. The English version of the questionnaire will be sent to English speakers and the Spanish version of the questionnaire will be sent to Spanish speakers. This aims to include a diverse sample of football staff from different regions, helping to better understand factors influencing adherence to movement guidelines and diet quality across various linguistic and cultural groups.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-16 (Actual)

PRIMARY OUTCOMES:
Moderate-to-Vigorous Physical Activity Time | From enrollment to the end of assessment
  Ratio scale, measured in minutes per week. From 0 minutes (low adherence) to 240+ minutes (high adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Light Physical Activity Time | From enrollment to the end of assessment
  Ratio scale, measured in hours per day. From 1 hours (low adherence) to 10+ hours (high adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Sedentary Time | From enrollment to the end of assessment
  Ratio scale, measured in hours per day. From 1 hour (high adherence) to 10+ hours (low adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Sleep Duration | From enrollment to the end of assessment
  Ratio scale, measured in hours per day. From 1 hours (low adherence) to 10+ hours (high adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Frequency of Fruit Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Do not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Vegetable Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Do not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Sweets Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 9 ("Do not eat it at all") to 0 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Whole Grain Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Do not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Diet Quality Summary Score | From enrollment to the end of assessment
  Accumulation of diet quality scores from Mini-Eat validated questions. A score of <61 is Unhealthy / Poor diet, a score between 60 and 68.9 is Intermediate / Diet needs improvement, a score of >69 is Healthy / Comparable to scores of >80.

SECONDARY OUTCOMES:
Strength Training Frequency | From enrollment to the end of assessment
  To determine whether participants do strength training exercises at least twice weekly. Nominal scale, with two possible values: Yes (high adherence) or No (low adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Sedentary Breaks | From enrollment to the end of assessment
  To identify whether participants interrupt prolonged sedentary periods. Nominal scale, with two possible values: Yes (high adherence) or No (low adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Screen Time Adherence | From enrollment to the end of assessment
  To evaluate whether participants limit daily recreational screen time to 3 hours or less. Nominal scale, with two possible values: Yes (high adherence) or No (low adherence).
  Question from the Whole Day Matters Toolkit: 24-hour movement questionnaire from The Canadian Society for Exercise Physiology.
Frequency of Legumes, Nuts, and Seeds Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Did not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Fish or Seafood Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Did not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Refined Grain Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 9 ("Did not eat it at all") to 0 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of High-Fat Dairy and Saturated Fats Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 9 ("Did not eat it at all") to 0 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.
Frequency of Low-Fat Dairy Intake | From enrollment to the end of assessment
  Ordinal scale. Scored from 0 ("Did not eat it at all") to 9 ("4 or more servings per day"). Question from validated Mini-Eat questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University Ramon Llull, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
* Information on adherence to the Canadian 24-hour Movement Guidelines, detailing, physical activity, sleep consistency, sedentary time, strength training, sedentary breaks, and screen time usage
  * Responses from the Mini-EAT dietary screening tool, detailing participants diet quality
  * Data related to participants job titles, gender, and location to assess correlations with physical movement and diet quality.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Lara-Breitinger KM, Medina Inojosa JR, Li Z, Kunzova S, Lerman A, Kopecky SL, Lopez-Jimenez F. Validation of a Brief Dietary Questionnaire for Use in Clinical Practice: Mini-EAT (Eating Assessment Tool). J Am Heart Assoc. 2023 Jan 3;12(1):e025064. doi: 10.1161/JAHA.121.025064. Epub 2022 Dec 30. PMID 36583423